CLINICAL TRIAL: NCT02305459
Title: CIRSE Registry for SIR-Spheres Therapy
Acronym: CIRT
Status: Completed | Type: Observational
Sponsor: Cardiovascular and Interventional Radiological Society of Europe (Other)
Responsible Party: Sponsor
Other Study IDs: CIRSECIRT
Record Dates: First submitted 2014-11-11; First posted 2014-12-02 (Estimated); Last update posted 2020-01-21 (Actual); Status verified 2020-01

CONDITIONS: Liver Carcinoma
Keywords: SIRT; microcatheter; primary liver tumor; secondary liver tumor; radioembolisation; QLQ-C30; CIRSE
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients treated with Radioembolisation: All Patients treated with Radioembolisation with yttrium-90 loaded SIR-Spheres microspheres are asked to be enrolled. In no way will participation in the registry influence the way in which the patient is treated or will it influence the quality of the treatment.
  In order to measure the palliative aspect of RE with SIR-Spheres microspheres, CIRT will incorporate a quality-of-life questionnaire. CIRT will be using EORTC's QLQ-C30 with the Hepatocellular carcinoma (HCC) Module to measure changes in the quality of life of the patient.
  Interventions: Device: Yttrium-90 loaded SIR-Spheres microspheres; Behavioral: QLQ-C30 with HCC module

INTERVENTIONS:
Device: Yttrium-90 loaded SIR-Spheres microspheres — Selective internal radiation therapy (SIRT), also called radioembolisation (RE), with SIR-Spheres microspheres is an endovascular procedure, included within the interventional oncologic technologies to treat primary and secondary liver tumours. Using a microcatheter, a precise dose of resin microspheres is released in the hepatic artery, where they are carried into the arterioles and selectively lodge in the tumour microvasculature. The microspheres are loaded with the radioactive yttrium-90, a high-energy beta-emitting isotope with a half-life of 64.1 hours. SIR-Spheres microspheres are manufactured by Sirtex Medical.
Behavioral: QLQ-C30 with HCC module — In order to measure the palliative aspect of RE with SIR-Spheres microspheres, CIRT will incorporate a quality-of-life questionnaire. CIRT will be using EORTC's QLQ-C30 with HCC Module to measure changes in the quality of life of the patient. The quality-of-life questionnaire will be offered to the patient before the treatment, shortly after the treatment (as soon as possible) and at every follow-up. Filling out the quality-of-life questionnaire is entirely voluntary for the patient.

SUMMARY:
The administration of SIR-Spheres microspheres (yttrium-90 resin microspheres) is a form of selective internal radiation therapy (SIRT) for the treatment of patients with primary and secondary liver tumours. The primary objective is to observe the real-life clinical application of radioembolisation with SIR-Spheres and the impact of the treatment in clinical practice. Secondary objectives are to observe safety and effectiveness of SIR-Spheres treatment in terms of adverse events, Overall Survival (OS), Progression-free survival (PFS), technical considerations, liver PFS and Quality of Life (QoL) + subgroup analyses

DETAILED DESCRIPTION:
Selective internal radiation therapy (SIRT), also called radioembolisation (RE), with SIR-Spheres microspheres is an endovascular procedure, included within the interventional oncologic technologies to treat primary and secondary liver tumours. Using a microcatheter, a precise dose of resin microspheres is released in the hepatic artery, where they are carried into the arterioles and selectively lodge in the tumour microvasculature. The microspheres are loaded with the radioactive yttrium-90, a high-energy beta-emitting isotope with a half-life of 64.1 hours. Following administration, 94% of the radiation is delivered in 11 days. Previous reports on the safety and efficacy of yttrium-90 resin microspheres for the treatment of primary and secondary liver tumours are very promising. In order to further improve the understanding of this therapy in its true clinical setting, the Cardiovascular and Interventional Radiological Society of Europe (CIRSE) initiated the CIRSE Registry for SIR-Spheres Therapy (CIRT), a phase 4 observational study that aims to collect robust data on the real-life clinical practice of radioembolisation with SIR-Spheres microspheres. Further, using the quality of life questionnaire QLQ-C30 with its hepatocellular carcinoma module (developed and verified by the European Organisation of Research and Treatment of Cancer (EORTC)), CIRT aims to collect data on the quality of life of patients treated with SIR-Spheres microspheres.

ELIGIBILITY:
Inclusion Criteria:

* Treatment of liver tumour with SIR-spheres microspheres
* Primary or secondary liver tumours
* Signed informed consent form
* 18 years or older

Exclusion criteria

* Under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients are only asked to be enrolled when they are treated with SIR-Spheres microspheres as part of the treatment determined by the treating clinician.
Sampling Method: Non-Probability Sample
Enrollment: 1051 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2020-01-01 (Actual)

PRIMARY OUTCOMES:
Description of the clinical context in which SIR-Spheres are applied | Baseline, follow-up every 3 months until 24 months
  Context of systemic therapy; intention of treatment; prior hepatic procedures; post hepatic procedures

SECONDARY OUTCOMES:
Adverse events | Every 3 months until 24 months
  Adverse events per follow-up
QLQ-C30 | Every 3 months until 24 months
  Quality of life using QLQ-C30 from baseline until 24 months
Overall survival | Every 3 months until 24 months
  Time till death
PFS | Every 3 months until 24 months
  Time to progression
Hepatic PFS | Every 3 months until 24 months
  Time to progression

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Helmberger, Prof, Principal Investigator — München Klinik Bogenhausen,Englschalkinger Str. 77, D-81925 München
Locations (1):
- Cardiovascular and Interventional Radiological Society of Europe, Vienna, Austria

REFERENCES:
- [Derived] Reimer P, Vilgrain V, Arnold D, Balli T, Golfieri R, Loffroy R, Mosconi C, Ronot M, Sengel C, Schaefer N, Maleux G, Munneke G, Peynircioglu B, Sangro B, Kaufmann N, Urdaniz M, Pereira H, de Jong N, Helmberger T. Factors Impacting Survival After Transarterial Radioembolization in Patients with Unresectable Intrahepatic Cholangiocarcinoma: A Combined Analysis of the Prospective CIRT Studies. Cardiovasc Intervent Radiol. 2024 Mar;47(3):310-324. doi: 10.1007/s00270-023-03657-x. Epub 2024 Feb 6. PMID 38321223
- [Derived] Kolligs F, Arnold D, Golfieri R, Pech M, Peynircioglu B, Pfammatter T, Ronot M, Sangro B, Schaefer N, Maleux G, Munneke G, Pereira H, Zeka B, de Jong N, Helmberger T; CIRT Principal Investigators. Factors impacting survival after transarterial radioembolization in patients with hepatocellular carcinoma: Results from the prospective CIRT study. JHEP Rep. 2022 Nov 25;5(2):100633. doi: 10.1016/j.jhepr.2022.100633. eCollection 2023 Feb. PMID 36593888
- [Derived] Helmberger T, Golfieri R, Pech M, Pfammatter T, Arnold D, Cianni R, Maleux G, Munneke G, Pellerin O, Peynircioglu B, Sangro B, Schaefer N, de Jong N, Bilbao JI; On behalf of the CIRT Steering Committee; On behalf of the CIRT Principal Investigators. Clinical Application of Trans-Arterial Radioembolization in Hepatic Malignancies in Europe: First Results from the Prospective Multicentre Observational Study CIRSE Registry for SIR-Spheres Therapy (CIRT). Cardiovasc Intervent Radiol. 2021 Jan;44(1):21-35. doi: 10.1007/s00270-020-02642-y. Epub 2020 Sep 21. PMID 32959085
- [Derived] Helmberger T, Arnold D, Bilbao JI, de Jong N, Maleux G, Nordlund A, Peynircioglu B, Sangro B, Sharma RA, Walk A. Clinical Application of Radioembolization in Hepatic Malignancies: Protocol for a Prospective Multicenter Observational Study. JMIR Res Protoc. 2020 Apr 22;9(4):e16296. doi: 10.2196/16296. PMID 32319960